CLINICAL TRIAL: NCT03605875
Title: Voicing Individual Concerns for Engagement in Hemodialysis (VOICE-HD): a Web Application for Rounds
Brief Title: A Web Application for Improving Communication on Hemodialysis Rounds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Stephanie Thompson, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00076483
Record Dates: First submitted 2018-07-18; First posted 2018-07-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Paper

STUDY DESIGN:
Intervention Model Description: 1:1 allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-App (Experimental): A customized web-app tool to be used by patients to communicate concerns to their nephrologist
  Interventions: Behavioral: Web-App
- Paper (Active Comparator): A customized paper tool to be used by patients to communicate concerns to their nephrologist
  Interventions: Behavioral: Paper

INTERVENTIONS:
Behavioral: Web-App — Cambian IT Health solutions from Surrey BC developed the infrastructure
  Arms: Web-App
Behavioral: Paper — Contains similar questions to the Web-App tool
  Arms: Paper

SUMMARY:
To evaluate a web application tool that hemodialysis patients can use outside of dialysis time to log and prioritize their concerns for the nephrologists. Specifically, the investigators will compare the usability of a web application tool to a structured paper form. The investigators will also use data from semi-structured interviews to better understand the experience and acceptability of the web app among patient participants randomized to the web application and among participating nephrologists.

Primary outcome

-Usability (effectiveness, efficiency, satisfaction)

Secondary outcomes

-Quality of the patient-physician interaction (Communication Assessment Tool (CAT-14))

DETAILED DESCRIPTION:
Usability is defined as Effectiveness (>70%)

* Number of people submitting a concern/ number of people with opportunity to submit a concern
* Number of concerns entered/number of times concern was satisfactorily addressed

Efficiency

* Proportion of non-completed tasks (<70%)
* The amount of time to complete one concern

Satisfaction

* Semistructured interviews
* Usability survey

ELIGIBILITY:
Inclusion Criteria:

* Chronic in-center hemodialysis patients in Edmonton, Alberta and Winnipeg, Manitoba
* Able to provide consent, understand and read English or have a family member that can do this for them

Exclusion Criteria:

* Planning to change modality within the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Effectiveness - Number of patients submitting a concern divided by the number of patients | 8 weeks
  Number of patients submitting a concern divided by the number of patients with an opportunity to submit a concern
Effectiveness - Number of concerns entered divided by the number of concerns that were satisfactorily addressed | 8 weeks
  Number of concerns entered divided by the number of concerns that were satisfactorily addressed
Efficiency - The amount of time to complete one concern | 8 weeks
  The amount of time to log a concern in the web app
Satisfaction - Usability survey | 8 weeks
  Usability survey Defined as greater than 70% of users who agree or strongly agree with the statement on the usability survey. Ranked on a 5 -point Likert scale

SECONDARY OUTCOMES:
Communication Assessment Tool | 8 weeks
  Items rated from 1 (poor) to 5 (excellent). Published at Makoul et al. Patient Educ Couns 2007

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Thompson, MD PhD, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - Edmonton General Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Seven Oaks General Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson S, Schick-Makaroff K, Bello A, Tonelli M, Wiebe N, Buzinski R, Courtney M, Szigety S, Shah N, Bohm C. Voicing Individual Concerns for Engagement in Hemodialysis (VOICE-HD): A Mixed Method, Randomized Pilot Trial of Digital Health in Dialysis Care Delivery. Can J Kidney Health Dis. 2021 Jul 27;8:20543581211032857. doi: 10.1177/20543581211032857. eCollection 2021. PMID 34377501